CLINICAL TRIAL: NCT02877914
Title: China Patient-centered Evaluative Assessment of Cardiac Events (PEACE): Retrospective Study of Patients With Heart Failure (HF)
Brief Title: China PEACE 5r-HF Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015BAI12B02-1
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure
Keywords: heart failure, retrospective
MeSH Terms: conditions — Heart Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational study — This is a non-interventional study, patients receive their usual treatment as determined by the physician.

SUMMARY:
This study will use a two-stage random sampling design to create a nationally representative sample of patients with heart failure (HF) in China. The investigators sought to describe the clinical profiles, to assess treatment patterns and in-hospital outcomes for HF, and to identify targets for care quality improvement.

DETAILED DESCRIPTION:
This study will use a two-stage random sampling design to create a nationally representative sample in China, and randomly sample patients with HF as a primary diagnosis, and were admitted to hospital from January 1st, 2015 to December 31st, 2015. The sample size is estimated to be 10,000.

The investigators will collect photocopies of the sampled medical records and centrally abstract detailed information, which included demographic characteristics, medical history, clinical features, diagnostic tests, in-hospital procedures, lab tests, treatments, and in-hospital outcomes. Data abstraction quality was monitored by random auditing of 5% of the medical records, with overall variable accuracy exceeding 98%.

Analyses will examine patient characteristics, diagnostic testing patterns, in-hospital treatments, in-hospital outcomes, and variation in results across regions and hospitals. Practical guidelines, quality evaluative system, and risk model will be established based on the findings, to improve patient outcomes for HF in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure as the primary reason for hospitalization, including both new-onset HF or decompensation of chronic HF。
* Hospitalized during January 1st, 2015 to December 31st, 2015
* Aged 18 years or above

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with primary reason for admission of heart failure, aged 18 years or above
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Death | Duration of hospitalization, an average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, MD, PhD, Principal Investigator — China National Center for Cardiovascular Disease; Harlan M Krumholz, MD, SM, Principal Investigator — Yale University
Locations (1):
- Zhengzhou People's Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu Y, Guan W, Masoudi FA, Wang B, He G, Spertus JA, Lu Y, Krumholz HM, Li J. Hospital Variation of Spironolactone Use in Patients Hospitalized for Heart Failure in China-The China PEACE Retrospective Heart Failure Study. J Am Heart Assoc. 2022 Oct 4;11(19):e026300. doi: 10.1161/JAHA.122.026300. Epub 2022 Sep 29. PMID 36172964
- [Derived] Yu Y, Gupta A, Wu C, Masoudi FA, Du X, Zhang J, Krumholz HM, Li J; China PEACE Collaborative Group. Characteristics, Management, and Outcomes of Patients Hospitalized for Heart Failure in China: The China PEACE Retrospective Heart Failure Study. J Am Heart Assoc. 2019 Sep 3;8(17):e012884. doi: 10.1161/JAHA.119.012884. Epub 2019 Aug 21. PMID 31431117
- [Derived] Yu Y, Spatz ES, Tan Q, Liu S, Lu Y, Masoudi FA, Schulz WL, Krumholz HM, Li J; China PEACE Collaborative Group. Traditional Chinese Medicine Use in the Treatment of Acute Heart Failure in Western Medicine Hospitals in China: Analysis From the China PEACE Retrospective Heart Failure Study. J Am Heart Assoc. 2019 Aug 6;8(15):e012776. doi: 10.1161/JAHA.119.012776. Epub 2019 Jul 31. PMID 31364457
- [Derived] Yu Y, Zhang H, Li X, Lu Y, Masoudi FA, Krumholz HM, Li J. The China Patient-centered Evaluative Assessment of Cardiac Events (China PEACE) retrospective heart failure study design. BMJ Open. 2018 May 10;8(5):e020918. doi: 10.1136/bmjopen-2017-020918. PMID 29748344